CLINICAL TRIAL: NCT03721848
Title: Impact of Health Promotion Interventions on the Management and Secondary Prevention of Non-Communicable Diseases Among Jordanians and Syrians in Jordan.
Brief Title: Impact of a Health and Mental Health Promotion Intervention Among Jordanians and Syrians.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Americares (Other); Royal Health Awareness Society (Unknown)
Responsible Party: Principal Investigator, Tara Powell, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17390
Record Dates: First submitted 2018-08-21; First posted 2018-10-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Mental Stress; Hypertension; Diabetes
MeSH Terms: conditions — Stress, Psychological; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: * Condition 1: an existing NCD preventive intervention consisting of 24 sessions, which are 45 minutes covering diabetes, hypertension, obesity, reproductive health, cardiovascular diseases, allergies and smoking;
  * Condition 2: The existing NCD preventive intervention with 4 added mental health awareness sessions covering traumatic stress reactions, individual strategies for coping with stress and traumatic events and collective strategies for coping with stress and trauma;
  * Condition 3: Treatment as usual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Community Clinic: NCD+MH (Experimental): The arm of this study consists of a 28 session intervention, which are 45 minutes and meet 2-3 times a month providing health awareness on non-communicable diseases diabetes, hypertension, obesity, reproductive health, cardiovascular diseases, allergies; smoking; traumatic stress reactions, individual strategies for coping with stress and traumatic events and collective strategies for coping with stress and trauma.
  Interventions: Behavioral: Healthy community clinic NCD+MH
- Healthy Community Clinic: NCD (Active Comparator): The arm of this study consists of a 24 session intervention, which are 45 minutes and meet 2 times a month providing health awareness on non-communicable disease diabetes, hypertension, obesity, reproductive health, cardiovascular diseases, allergies; smoking.
  Interventions: Behavioral: Healthy community clinic NCD
- Treatment as usual (No Intervention): This is treatment as usual where there is no intervention, but patients attend the clinic for treatment of non-communicable diseases.

INTERVENTIONS:
Behavioral: Healthy community clinic NCD+MH — NCD+MH Awareness Intervention Overview:
  i. Patients are assigned, at minimum, one health awareness lecture per month with a total of 28 lectures possible ii. Patients attend lectures on specific topics given by MoH staff, mainly nurses.
  iii. Topics tackled include: Diabetes, Hypertension, Asthma, Cardiovascular Disease, Reproductive Health, Healthy Nutrition, Smoking, Emotional Wellness, Stress Relief and Positive Coping.
  iv. Group nutrition and physical fitness counselling are incorporated into most health awareness lectures
  Arms: Healthy Community Clinic: NCD+MH
Behavioral: Healthy community clinic NCD — i. Patients are assigned, at minimum, one health awareness lecture per month with a total of 24 lectures possible ii. Patients attend lectures on specific topics given by MoH staff, mainly nurses.
  iii. Topics tackled include: Diabetes, Hypertension, Asthma, Cardiovascular Disease, Reproductive Health, Healthy Nutrition, and Smoking iv. Group nutrition and physical fitness counselling are incorporated into most health awareness lectures
  Arms: Healthy Community Clinic: NCD

SUMMARY:
Given the heightened risk of NCDs and mental health issues, it is critical for Jordanians and Syrian refugees to have access to prevention based health services. To address this need, the following project seeks to examine the capacity of Primary Care Health Centers to provide preventive services to empower patients to manage NCDs and potential mental health issues for those who are experiencing distress.

The primary research question in this evaluation study is:

Does prevention-based health and mental health services in primary health clinics improve health status of Jordanians and Syrian refugees?

This research proposal will consist of three study conditions examining:

* Condition 1: an existing NCD preventive intervention consisting of 24 sessions, which are 45 minutes covering diabetes, hypertension, obesity, reproductive health, cardiovascular diseases, allergies and smoking;
* Condition 2: The existing NCD preventive intervention with 4 added mental health awareness sessions covering traumatic stress reactions, individual strategies for coping with stress and traumatic events and collective strategies for coping with stress and trauma;
* Condition 3: Treatment as usual

A group randomized study will be conducted in three clinics with patients of the respective clinics. The clinics will be identified prior to the study based on similar demographics, service utilization and staff capacity. Once the three clinics are identified they will be selected to one of the three study conditions. This research will be conducted in collaboration with the University of Illinois (UIUC), AmeriCares, and the Royal Health Awareness Society (RHAS) of Jordan. AmeriCares will work as the operational humanitarian organization collaborating with and providing support to RHAS and UIUC. RHAS's healthy community clinic is a community-based health project launched in 2011 conducted with the Ministry of Health (MOH). The project aims to build the capacity of participating Health Centers to provide better preventative services to empower patients to manage their diseases and reduce future complications. The Healthy Community Clinic, established within existing MOH facilities, provides medical practitioners with the training and resources necessary to implement management and prevention-based care to patients in underserved communities.

ELIGIBILITY:
Inclusion Criteria:Eligible patients are referred to the study through the treating MOH physicians at the health centers. Through an initial screening process, patients will be assessed for eligibility via inclusion/exclusion criteria by trained nurses. As stated, the nurses will be trained in the data collection procedures by the Research Manager and potential subjects will be fully informed that they can still receive health care services even if they have no interest in participating in the research. This information will be received through the patient information and self-report.

1. Inclusion Criteria (at least two of the following):

   * Obesity, defined as BMI ≥ 30
   * Fasting blood glucose ≥ 100 ml/dl
   * Systolic blood pressure ≥ 120 mmHg and/or diastolic blood pressure ≥ 80 mmHg
   * Self-reported uncontrolled dyslipidaemia, cholesterol >240, LDL >190, HDL < 40 ad/or TG >500
   * Asthma
   * Diabetes
   * Hypertension

   Exclusion Criteria:
2. Exclusion criteria:

   * Renal dysfunction: also known as renal insufficiency or renal failure; assessed by self-report
   * Heart failure: also known as congestive heart disease or chronic heart failure; assessed by self-report
   * Functional disability: defined as any long-term activity limitation due to disease or injury; assessed by self-report
   * Liver dysfunction: also known as liver failure, acute or chronic; assessed by self-report
   * Uncontrolled Resistant Hypertension: defined as blood pressure remaining above the threshold despite lifestyle modifications and concurrent use of at least three antihypertensive medications from different classes with one being a diuretic10-11assessed by self-report
   * Pregnant women
   * Uncontrolled Hypothyroidism * Pregnant women are excluded because it would be almost impossible to find any reduction in pregnant women weight and that will show a negative impact of HCC intervention on weight reduction. Therefore, inclusion of pregnant women could be a confounding factor to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Health Behavior-Fruit Intake frequency (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Likert 5 point question assessing frequency of fruit intake within a week (a. none, b. 1-2 times per week, c. 3-4 times per week, d. 5 + times per week.
Health Behavior-Vegetable Intake (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Likert 5 point question assessing frequency of vegetable intake within a week (a. none, b. 1-2 times per week, c. 3-4 times per week, d. 5 + times per week.
Health Behavior-Bread Intake (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Likert 5 point question assessing frequency of bread intake within a week (a. none, b. 1-2 times per week, c. 3-4 times per week, d. 5 + times per week.
Incidence of Smoking (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Yes/no question asking participants if they smoke. If they answer yet to smoking they are prompted to ask how many cigarettes per week.
Health Behavior- Level of Physical Activity (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Question inquiring how much physical activity participants get per week. Likert question Ranging from a. 30 minutes b.30 min to 1 hour c. 1-2 hours, d. 2-5 hours, e. more than 5 hours
Health Behavior-Amount of Red Meat Intake (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Likert 5 point question assessing frequency of red meat intake within a week (a. none, b. 1-2 times per week, c. 3-4 times per week, d. 5 + times per week.

SECONDARY OUTCOMES:
Duke Health Profile (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Duke Health Profile: 17-item standardized self-report instrument containing six health measures (physical, mental, social, general, perceived health, and self-esteem), and four dysfunction measures (anxiety, depression, pain, and disability).
Blood Pressure (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Trained nurses will collect Blood Pressure: Patients will be asked to remain seated with their legs uncrossed for at least 5 minutes before blood pressure measurements can be taken. In a seated position, systolic and diastolic blood pressure will be measured in mmHg by sphygmomanometer. This measurement should be repeated three times and the average of the second and third measurements should be calculated for data analysis.
BMI (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Patients should be asked to remove their shoes and any outer garments, while maintaining cultural respect. Calibrated scales will be used to measure body weight to the nearest 0.5 kg. Height will be measured to the nearest 0.1 cm using the height rod attached to the scale.23The BMI will be calculated by dividing the mass in Kg over the square of the height in meters according to the equation below:
  BMI = Mass (kg)/Height (m2)
Laboratory tests: fasting blood glucose (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Appointments for laboratory tests will occur in the mornings to allow for patients to fast overnight (a minimum of 8 hours). MedLabs phlebotomists will collect the samples. The amount of blood to be collected is 3 ml. Each tube is clearly marked with the volume of blood to be collected. Any specimen not meeting the test requirement in terms of volume must be rejected.
Laboratory tests: HbA1c (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Appointments for laboratory tests will occur in the mornings to allow for patients to fast overnight (a minimum of 8 hours). MedLabs phlebotomists will collect the samples. The amount of blood to be collected is 3 ml. Each tube is clearly marked with the volume of blood to be collected. Any specimen not meeting the test requirement in terms of volume must be rejected.
Laboratory tests: total cholesterol (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Appointments for laboratory tests will occur in the mornings to allow for patients to fast overnight (a minimum of 8 hours). The amount of blood to be collected is 3 ml. Each tube is clearly marked with the volume of blood to be collected. Any specimen not meeting the test requirement in terms of volume must be rejected.
Health Behavior (Hypertension, Diabetes, Mental health, Nutrition) Knowledge Survey (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  22 item questionnaire developed to measure knowledge of risk and management of: hypertension, diabetes, mental health, nutrition. Participant can report yes/no/I don't know to each question. The correct items will then be summed to identify the levels of knowledge change across time.
Brief Trauma Questionnaire (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Brief Trauma Questionnaire:
  The BTQ is a 10 item self-report questionnaire derived from the Brief Trauma Interview.
Primary Care PTSD (Assessing Change) | Baseline, Six Months, 12 Months, 18 months
  Six item screen derived from the PTSD Checklist-Civilian Version to help primary care settings screen for persons with possible PTSD symptoms. The five point Likert Scale ranges from not at all to extremely inquiring on prevalence of PTSD symptoms (e.g. had repeated disturbing memories about an event; c) Avoided activities or situations because they reminded you of a stressful experience)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Powell, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Royal health Awareness Society, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Powell TM, Shin OJ, Li SJ, Hsiao Y. Post-traumatic stress, social, and physical health: A mediation and moderation analysis of Syrian refugees and Jordanians in a border community. PLoS One. 2020 Oct 23;15(10):e0241036. doi: 10.1371/journal.pone.0241036. eCollection 2020. PMID 33095832